CLINICAL TRIAL: NCT00202826
Title: Parapneumonic Effusion in Children Study
Brief Title: Study of Fluid Collection of the Chest in Children With Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Helen DeVos Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-181
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2009-01

CONDITIONS: Community Acquired Bacterial Pneumonia; Paraneumonic Effusion
MeSH Terms: interventions — Drainage

INTERVENTIONS:
Procedure: Video Assisted Thorascopic Surgery Thoracostomy Tube Placement & Drainage

SUMMARY:
The purpose of this study is to determine the best treatment for children with a fluid collection in the chest associated with an underlying pneumonia. Researchers generally agree that a child with a large fluid collection in the chest need to have the fluid drained in addition to anitbiotics. There have been many treatments studied in children that have been shown to be effective and safe, but the treatments have never been compared to each other in a randomized controlled study.

The optimal treatment of pediatric parapneumonic effusions remains controversial. The objective of this study is to compare the use of conventional management (antibiotics with thoracostomy tube placement) with primary thorascopic drainage (see protocol). Our hypothesis is that pediatric patients with parapneumonic effusion, regardless of pleural fluid composition and loculations, have decreased morbidity when treated with early thoroscopic adhesiolysis (VATS) compared with conservative treatment.

DETAILED DESCRIPTION:
The ultimate objective of this study is to rationalize treatment decisions. It is our hope that this pilot study will provide the basis for further randomized prospective studies. The expected benefit is that the current treatment and outcome of pediatric parapneumonic effusions will be determined. Insights into the therapy that results in the least morbidity, hospital days, (and therefore cost) will be elucidated. If our hypothesis is valid, then a more aggressive surgical approach to the treatment of a parapneumonic effusion may be warranted. If the hypothesis is not valid, then the appropriate treatment for a parapneumonic effusion, irrespective of institution and personal opinion, should become more apparent.

ELIGIBILITY:
Inclusion Criteria:

1. consecutive pediatric patients with a bacterial pneumonia and parapneumonic effusion
2. community acquired disease
3. children age 0 to 18 years

Exclusion Criteria:

1. hospital acquired pneumonia
2. thoracentesis or chest tube drainage outside hospital
3. patients with incorrected cardiac disease

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2003-11; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
establish morbidity outcomes
duration of fever
number of procedures
days with a chest drainage device
total hospital days

SECONDARY OUTCOMES:
Days of oxygen requirement
Days of narcotic use
Complication rate
Number of radiographic procedures

CONTACTS AND LOCATIONS:
Overall Officials: John Winters, MD, Principal Investigator — Helen DeVos Children's Hospital
Locations (1):
- DeVos Children's Hospital, Grand Rapids, Michigan, United States